CLINICAL TRIAL: NCT03143998
Title: A Multi-Site, Open-Label, Trial of the Efficacy and Safety of Fixed-dose Elbasvir/Grazoprevir (EBR/GZR) in Brazilian Patients With Chronic Hepatitis C Virus (HCV) Genotype 1 Infection With Advanced Fibrosis (F3 and F4)
Brief Title: Efficacy and Safety of Elbasvir/Grazoprevir in Brazilian Participants With Chronic Hepatitis C Virus (HCV) Genotype 1 Infection With Advanced Fibrosis (F3 and F4)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-089
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HCV GT1a TN (Experimental): Participants with HCV GT1a infection who are TN will take MK-5172A for 12 weeks.
  Interventions: Drug: MK-5172A
- HCV GT1a TE (Experimental): Participants with HCV GT1a infection who are TE will take MK-5172A for 12 weeks.
  Interventions: Drug: MK-5172A
- HCV GT1b TN (Experimental): Participants with HCV GT1b infection who are TN will take MK-5172A for 12 weeks.
  Interventions: Drug: MK-5172A
- HCV GT1b TE (Experimental): Participants with HCV GT1b infection who are TE will take MK-5172A for 12 weeks.
  Interventions: Drug: MK-5172A

INTERVENTIONS:
Drug: MK-5172A — A single FDC tablet containing grazoprevir 100 mg + elbasvir 50 mg taken once daily by mouth.
  Other Names: ZEPATIER®

SUMMARY:
This is a non-randomized, open-label study of a fixed dose combination (FDC) of elbasvir (50 mg) and grazoprevir (100 mg) (EBR/GZR or MK-5172A) in participants with chronic hepatitis C virus (HCV) genotype 1 (GT1) infection with advanced fibrosis with and without human immunodeficiency virus (HIV) co-infection. All participants will be either HCV treatment naïve (TN) or treatment experienced (TE).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) male and female participants with chronic HCV GT1 infection who reside in Brazil
* HCV RNA (≥ 10,000 IU/mL in peripheral blood) at the time of screening
* Has documented chronic HCV GT1 (1a; 1b) infection (with no evidence of non-typeable or mixed genotype) infection.

  * positive for anti HCV antibody, HCV RNA, or HCV GT1 at least 6 months before screening, or
  * positive for anti-HCV antibody or HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of chronic hepatitis C (CHC) disease, such as the presence of fibrosis)
* Is otherwise healthy as determined by the medical history, physical examination, and clinical laboratory measurements at the time of screening
* Has a history of advanced fibrosis (F3 or F4) as follows:

  * F4: FibroSure®/APRI + FibroTest®
  * Liver biopsy result of METAVIR stage 3 or 4 fibrosis (or its grading system equivalency to advanced fibrosis)
  * FibroScan® result > 9.5 kPa (F3 or F4)
* Has liver imaging within 6 months of Day 1 (start of treatment) with no evidence of hepatocellular carcinoma (HCC)
* Is TN or TE
* Is a male, is a female who is not of reproductive potential, or is a female of reproductive potential who agrees to avoid becoming pregnant from Day 1 (start of treatment) through 14 days after the last dose of study drug (or longer if dictated by local regulations)
* For HIV-infected participants, has HIV-1 infection documented prior to screening, and is either not currently on antiretroviral therapy (ART) and has no plans to initiate ART or has well-controlled HIV on ART as per study criteria

Exclusion Criteria:

* Has prior treatment with direct acting antiviral (DAA) therapy with the exception of boceprevir, telaprevir, and simeprevir
* Has evidence of decompensated liver disease as manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy, or other signs or symptoms of active advanced liver disease
* Is classified as Child-Pugh B or C or has a Child-Pugh-Turcotte score > 6
* Is hepatitis B surface antigen (HBsAg) positive at screening
* Is under evaluation for HCC or other active or suspected malignancy
* Is currently participating or has participated in a study with an investigational compound within 1 year of signing informed consent and is not willing to refrain from participating in another such study during the course of this study
* Has clinically-relevant drug or alcohol abuse within 12 months of screening
* Is a female and is pregnant or breastfeeding, or expecting to conceive or donate eggs from Day 1 (start of treatment) through 14 days after the last dose of study drug or longer if dictated by local regulations; or is a male participant who is expecting to donate sperm from Day 1 (start of treatment) through 14 days after the last dose of study drug or longer if dictated by local regulations
* Has any clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with treatment, assessment or compliance with the protocol or any medical/surgical conditions that may result in a need for hospitalization during the period of the study; or is currently under evaluation for a potentially clinically-significant illness (other than HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-12 (Estimated); Primary Completion 2019-01-12 (Estimated); Study Completion 2019-01-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving sustained virologic response (SVR) 12 weeks after the end of all study therapy (SVR12) | Week 24 (12 weeks after completing study therapy)
  SVR12 will be declared when a participant has HCV ribonucleic acid (RNA) < lower limit of quantification (LLOQ) 12 weeks after the end of all study therapy. Levels of HCV RNA will be determined with the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test, v2.0, which has a LLoQ of 15 IU/mL.
Percentage of participants experiencing an adverse event (AE) | Up to 14 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Percentage of participants withdrawing from study therapy due to an AE | Up to 12 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of participants achieving SVR 24 weeks after the end of all study therapy (SVR24) | Week 36 (24 weeks after completing study therapy)
  SVR24 will be declared when a participant has HCV RNA < LLOQ 24 weeks after the end of all study therapy. Levels of HCV RNA will be determined with the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test, v2.0, which has a LLoQ of 15 IU/mL.
Emergence of viral resistance-associated variants (RAVs) | Up to 12 weeks
  The RAVs resistant to EBR or GZR, including the association of baseline RAVs with treatment outcomes (SVR12 and SVR24) and the emergence of RAVs in participants who fail to achieve SVR will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Undecided